CLINICAL TRIAL: NCT05305287
Title: Quantitation of Hepatic Mitochondrial Fluxes in Humans With Nonalcoholic Fatty Liver Disease (NAFLD)
Brief Title: Quantifying Hepatic Mitochondrial Fluxes in Humans
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Luke Norton, Assistant Professor, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: HSC20210284H; 1R01DK129676-01A1 (NIH)
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Type 2 Diabetes; Mitochondrial Metabolism Disorders
Keywords: NAFLD; Diet; Exercise
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus, Type 2; Motor Activity | interventions — Pioglitazone

STUDY DESIGN:
Intervention Model Description: Patients with T2D and NAFL or NASH will be randomly assigned to receive placebo or pioglitazone treatment groups.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- NAFL TZD (Experimental): T2D with non-alcoholic fatty liver (NAFL), treated with pioglitazone
  Interventions: Drug: Pioglitazone
- NAFL Placebo (Placebo Comparator): T2D with non-alcoholic fatty liver (NAFL), treated with placebo
  Interventions: Other: Placebo
- NASH TZD (Experimental): T2D with non-alcoholic steatohepatitis (NASH), treated with pioglitazone
  Interventions: Drug: Pioglitazone
- NASH Placebo (Placebo Comparator): T2D with non-alcoholic steatohepatitis (NASH), treated with placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Pioglitazone — An insulin sensitizer and anti-diabetic agent. Participants will be started on 15 mg/day, increased to 30 mg/day at week 2 and then to 45 mg/day at week 4.
  Other Names: Actos
  Arms: NAFL TZD; NASH TZD
Other: Placebo — Placebo for pioglitazone
  Arms: NAFL Placebo; NASH Placebo

SUMMARY:
In this study the investigators will quantitate hepatic mitochondrial fluxes in T2D patients with NAFL and NASH before and after 16-weeks treatment with the insulin sensitizer pioglitazone

DETAILED DESCRIPTION:
The study team will examine hepatic mitochondrial TCA flux and pyruvate cycling (oral [U-13C]-propionate), hepatic gluconeogenesis (oral 2H2O), and hepatic insulin sensitivity (intravenous [3,4-13C2]-glucose with euglycemic insulin clamp) before and after 16 weeks treatment with the FDA approved insulin sensitizer pioglitazone. These studies will be performed in (i) type 2 diabetic subjects with NAFL but without evidence of fibrosis, and (ii) type 2 diabetic patients with NASH. Liver biopsies will be obtained before and after treatment for the diagnosis of NAFL/NASH and for molecular analyses.

ELIGIBILITY:
T2D with NAFL

Inclusion Criteria:

* Confirmed T2D based on OGTT (2 h glucose ≥200 mg/dl).
* Treated with diet, metformin, and/or sulfonylurea and in good general health determined by medical history, physical exam, and routine blood chemistries;
* age = 18-80 years;
* BMI = 25-40 kg/m2;
* HbA1c = 7-10%; stable body weight (±4 pounds) over the preceding 3-months;
* not taking any medication known to affect glucose metabolism other than antidiabetic medications.
* Evidence of moderate/severe fatty liver (steatosis; grade S2/S3 on FibroScan corresponding to ≥10% fat on MRI-PDFF) and no/minimal hepatic fibrosis (grade F0/F1 on FibroScan).

Exclusion Criteria:

* Alcohol consumption >14 units/week for women and >21 units/week for men.
* Cirrhosis (fibrosis stage 4).
* Type 1 diabetes and/or GAD positive subjects.
* Subjects not drug naive or have been on metformin more than 3 months.
* Presence of proliferative retinopathy.
* Urine albumin excretion > 300 mg/day.
* Evidence of other forms of chronic liver disease, including alcoholic liver disease, hepatitis B and C, primary biliary cholangitis, suspected/proven liver cancer and any other liver disease other than NAFLD.
* History of NY Class III-IV heart failure

T2D with NASH

Inclusion Criteria:

* Confirmed T2D based on OGTT (2 h glucose ≥200 mg/dl).
* Treated with diet, metformin, and/or sulfonylurea and in good general health determined by medical history, physical exam, and routine blood chemistries;
* age = 18-80 years;
* BMI = 25-40 kg/m2;
* HbA1c = 7-10%;
* stable body weight (±4 pounds) over the preceding 3-months;
* not taking any medication known to affect glucose metabolism other than antidiabetic medications.
* Evidence of moderate/severe fatty liver (steatosis; grade S2/S3 on FibroScan corresponding to ≥10% liver fat on MRI-PDFF) and moderate/severe hepatic fibrosis (grade F2/F3 on FibroScan).

Exclusion Criteria:

* Alcohol consumption >14 units/week for women and >21 units/week for men.
* Cirrhosis (fibrosis stage 4).
* Type 1 diabetes and/or GAD positive subjects.
* Subjects not drug naive or have been on metformin more than 3 months.
* Presence of proliferative retinopathy.
* Urine albumin excretion > 300 mg/day.
* Evidence of other forms of chronic liver disease, including alcoholic liver disease, hepatitis B and C, primary biliary cholangitis, suspected/proven liver cancer and any other liver disease other than NAFLD.
* History of NY Class III-IV heart failure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Effect of pioglitazone on hepatic mitochondrial TCA cycle fluxes | Baseline, week 16
  Quantitated using a combine stable isotope approach before and after treatment with pioglitazone

SECONDARY OUTCOMES:
Mean absolute change from baseline in liver fat content by magnetic resonance Imaging - Proton Density Fat Fraction (MRI-PDFF) | Baseline, Week 16
  Mean absolute change from baseline in liver fat content by MRI-PDFF
Mean change from baseline in body weight | Baseline, Week 16
  Mean change from baseline in body weight
Mean change from baseline in body composition | Baseline, Week 16
  Mean change from baseline in lean and fat mass measured by DEXA
Quantitate the effect of pioglitazone on liver histology by improvement of fibrosis | Week 16
  Percentage of Participants with ≥1 Point Decrease in Fibrosis Stage with No Worsening of NASH on Liver Histology
Quantitate the effect of pioglitazone on NAFLD Activity Score (NAS) | Week 16
  Percentage of Participants that Achieve a ≥2 Point Decrease in NAS on Liver Histology, with ≥1 Point Reduction in at Least 2 NAS Components
Examine the effect of pioglitazone on non-invasive markers of NAFLD | Baseline, Week 16
  Mean change from baseline in Fibrosis-4 (FIB-4), transient elastography (Fibroscan®), NAFLD fibrosis score (NFS), alanine transaminase (ALT) and aspartate transaminase (AST)
Effect of pioglitazone on the hepatic lipidome | Baseline, Week 16
  Lipidomics will be carried out using mass-spectrometry methods
Effect of pioglitazone on hepatic gene regulatory networks | Baseline, Week 16
  Multimodal RNA-Seq and ATAC-Seq will be used to examine gene regulatory networks in liver samples

CONTACTS AND LOCATIONS:
Overall Officials: Luke Norton, PhD, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (2):
- United States (2):
  - Texas Diabetes Institute - University Health System, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas